CLINICAL TRIAL: NCT05863403
Title: Effect of Neuromuscular Training Versus Traditional Exercise on Balance and Fall in Geriatric Population With Fall Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/529
Record Dates: First submitted 2023-03-18; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Geriatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training (Experimental)
  Interventions: Diagnostic Test: Neuromuscular Training
- Traditional Exercise (Active Comparator)
  Interventions: Diagnostic Test: Traditional Exercise

INTERVENTIONS:
Diagnostic Test: Neuromuscular Training — Neuromuscular Training on Balance and Fall in Geriatric Population With Fall Risk
  Arms: Neuromuscular Training
Diagnostic Test: Traditional Exercise — Traditional Exercise on Balance and Fall in Geriatric Population With Fall Risk
  Arms: Traditional Exercise

SUMMARY:
To determine the effect of neuromuscular training versus traditional exercise on balance and fall in geriatric population with fall risk

DETAILED DESCRIPTION:
neuromuscular training versus traditional exercise for the balance messurement of fall population with geriatric

ELIGIBILITY:
Inclusion Criteria:

* Patients with balance and fall problem doing physical therapy with an age over 60 years old and willing to participate will be included in the study.

Exclusion Criteria:

* Patient with other serious comorbidities and suffering from heart or kidney disease will not be include or unwilling to participate and those who will aged under 60 years will be excluded from the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale and Falls Efficiancy Scale international | 6 Month
  FES and BFalls Efficiancy Scale international the balance for Geriatric Population With Fall Risk

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudhary Muhammad Akram Teaching and research hospital, Jinnah Hospital Lahore and Mayo Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No